CLINICAL TRIAL: NCT03305783
Title: The Influence of Cholecystectomy on Secretion of Incretin Hormones
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Henriette Holst Nerild, MD, Ph.D. student, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-15016324
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — biopsies from the gallbladder and ductus cysticus after cholecystectomy biopsies only collected from 12 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients having cholecystectomy: Healthy, normal weight patients (BMI<27) undergoing elective cholecystectomy will have a meal test performed before and after surgery.
  Interventions: Procedure: cholecystectomy
- Healthy controls: Healthy matched controls will have one meal test performed.

INTERVENTIONS:
Procedure: cholecystectomy — elective cholecystectomy performed due to gallstones, cholecystitis or other non-malignant conditions and therefore done regardless of the protocol of this study.
  Groups: Patients having cholecystectomy

SUMMARY:
The effect of cholecystectomy on postprandial plasma GLP-1 responses (primary endpoint) and glucose metabolism will be evaluated in 30 patients planned to undergo elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
This is an observational, parallel-group study in 30 patients with gallstone disease and 10 healthy control subjects. In patients undergoing cholecystectomy a 4h-meal test (liquid mixed meal) will be conducted at baseline (1-2 weeks before surgery) and again within 4 weeks after the cholecystectomy. Healthy subjects will be submitted to a single 4h-meal test.

Secondary endpoints include changes in plasma glucose, insulin, glucagon, GIP, PYY, gastrin, CCK, fibroblast growth factor 19 (FGF-19) and bile acids. Furthermore, secondary endpoints include changes in gastric emptying (evaluated by the paracetamol method).

ELIGIBILITY:
Inclusion Criteria:

* caucasians above 18 years of age, having an elective cholecystectomy performed because of gallstone disease.
* normal fasting plasma glucose and HbA1c
* normal hgb
* Normal gallbladder ejection fraction

Exclusion Criteria:

* liver disease
* kidney disease
* diabetes
* ongoing infection
* abdominal pain not related to gall stones
* BMI <18,5 kg/m2 eller BMI >30 kg/m2
* prior abdominal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A healthy, normal weight population undergoing elective surgery because of gall stone disease.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Postprandial GLP-1 response | 240 min
  Gut derived hormone secretion after a 4 h meal test measured in pmol/liter

SECONDARY OUTCOMES:
plasma glucose | 240 min
  measured in mmol/liter
gastric emptying | 240 min
  evaluated by the paracetamol method
Resting metabolic rate | 240 min
  evaluated by calorimetry
insulin | 240 min
  measured in pmol/liter
Glucagon | 240 min
  measured in pmol/liter
PYY | 240 min
  peptide YY, measured in pmol/liter
GIP | 240 min
  measured in pmol/liter
CCK | 240 min
  Cholecystokinin, measured in pmol/liter
FGF-19 | 240 min
  Fibroblast growth factor 19, measured in ng/mL
Gastrin | 240 min
  measured in pmol/liter
Bile acids | 240 min
  measured in nmol/ml

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD. Proff., Study Director — Center for Clinical Metabolic Research, Gentofte hospital
Locations (1):
- Center for Clinical Metabolic Research, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No